CLINICAL TRIAL: NCT02493673
Title: The Effects of Continuous Positive Airway Pressure Therapy Withdrawal on Cerebral Vascular Reactivity and Brain Oxygenation in Patients With Obstructive Sleep Apnoea: A Randomised Controlled Trial
Brief Title: The Effects of CPAP Withdrawal on Cerebral Vascular Reactivity and Brain Oxygenation in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KEK-ZH-Nr. 2014-0684
Record Dates: First submitted 2015-06-30; First posted 2015-07-09 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continuous Positive Airway Pressure; Stroke; Cerebrovascular reactivity; Brain oxygenation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- CPAP therapy (Active Comparator): Continuous positive airway pressure therapy
  Interventions: Device: Continuous positive airway pressure device
- Sham CPAP (Sham Comparator): Sham- Continuous positive airway pressure
  Interventions: Device: Continuous positive airway pressure device

INTERVENTIONS:
Device: Continuous positive airway pressure device — (ResMed Spirit S8)

SUMMARY:
Obstructive sleep apnoea (OSA) is a highly prevalent sleep-related breathing disorder associated with adverse cardiovascular outcome. Underlying mechanisms are subject of debate. A causal relationship between OSA and systemic hypertension as well as peripheral endothelial dysfunction was shown, and there is accumulating evidence from physiologic and observational studies that cerebral autoregulation is insufficient to protect the brain from the nocturnal consequences of OSA. However, there are no data from randomised controlled trials proving a causal relationship between OSA and impaired cerebral vascular reactivity (CVR). The aim of this randomised controlled trial is to study the effects of a short-term CPAP withdrawal, and thus returning OSA, on daytime CVR and brain oxygenation to establish whether there is a causal relationship between OSA and cerebral vascular damage.

ELIGIBILITY:
Inclusion Criteria:

* Objectively confirmed OSA (at the time of original diagnosis) with an oxygen desaturation index (ODI) and apnoea-hypopnoea-index (AHI) of ≥20/h.
* Currently an oxygen desaturation index (≥4% dips) of ≥15/h during an ambulatory nocturnal pulse oximetry performed on the last night of a four-night period off CPAP.
* Treated with CPAP for more than 12 months
* Device usage >4h per night, >80% of the last 365 days, and AHI<10 with treatment (according to CPAP machine download data).
* Age between 20 and 75 years.
* Written informed consent as documented by signature.

Exclusion Criteria:

* Previous ischemic or haemorrhagic stroke; known cerebral aneurysm or arterio-venous malformation.
* Carotid artery stenosis > 70%
* Use of alpha- and beta-adrenergic blocking medication, antianginal medications, triptans, selective COX-inhibitors
* Unstable, untreated coronary or peripheral artery disease, severe arterial hypertension or hypotension (>180/110 or <90/60mmHg)
* Implanted pacemaker or internal cardiac defibrillator
* Changes in medication during the trial
* Previous ventilatory failure (awake SpO2 <93% andPaCO2>6kPa).
* Obesity hypoventilation syndrome, COPD
* Previously diagnosed with Cheyne-Stokes breathing.
* Current professional driver or any previous sleep related driving accidents.
* Caffeine or nicotine abuse 12 hours before measurements

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular reactivity (CVR) | Change from baseline in CVR after 2 weeks of CPAP withdrawal
  CVR measured non-invasively by blood oxygen level-dependent (BOLD) magnetic resonance imaging (MRI) under controlled cardiovascular reactivity stimulation during wakefulness

SECONDARY OUTCOMES:
Ambulatory morning blood pressure | Change from baseline in ambulatory morning blood pressure after 2 weeks of CPAP withdrawal
Resting heart rate | Change from baseline in resting heart rate after 2 weeks of CPAP withdrawal
Apnoea-hypopnoea-index (AHI) | Change from baseline in AHI after 2 weeks of CPAP withdrawal
Oxygen Desaturation Index (ODI) | Change from baseline in ODI after 2 weeks of CPAP withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Principal Investigator — University of Zurich
Locations (1):
- Pulmonary Division, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Thiel S, Gaisl T, Lettau F, Boss A, Winklhofer S, Kohler M, Rossi C. Impact of hypertension on cerebral microvascular structure in CPAP-treated obstructive sleep apnoea patients: a diffusion magnetic resonance imaging study. Neuroradiology. 2019 Dec;61(12):1437-1445. doi: 10.1007/s00234-019-02292-z. Epub 2019 Sep 16. PMID 31529145
- [Derived] Thiel S, Haile SR, Peitzsch M, Schwarz EI, Sievi NA, Kurth S, Beuschlein F, Kohler M, Gaisl T. Endocrine responses during CPAP withdrawal in obstructive sleep apnoea: data from two randomised controlled trials. Thorax. 2019 Nov;74(11):1102-1105. doi: 10.1136/thoraxjnl-2019-213522. Epub 2019 Aug 29. PMID 31467191